CLINICAL TRIAL: NCT00142389
Title: Comparison of Maternal and Infant Immunization Strategies to Prevent Pneumococcal Disease
Brief Title: Mother's Gift Project
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Thrasher Research Fund (Other); Bill and Melinda Gates Foundation (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Wyeth is now a wholly owned subsidiary of Pfizer (Industry); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 26748
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2005-08

CONDITIONS: Pneumococcal Infections
Keywords: gestational immunization,; infant antibody,; cord antibody
MeSH Terms: conditions — Pneumococcal Infections

INTERVENTIONS:
Biological: pneumococcal polysaccharide and protein conjugate vaccines

SUMMARY:
This prospective randomized evaluation of pneumococcal vaccine immunization of pregnant mothers, followed by pneumococcal conjugate immunization of their children is designed to assess the effects of these strategies on the immunogenicity and safety of both vaccines. We hypothesize that maternal followed by infant immunization will be safe and will provide higher levels of antibody from birth through 12 months of age.

DETAILED DESCRIPTION:
This is a randomized vaccine evaluation in 4 groups of mothers and their infants, to assess the effect of maternal immunization on the infants' response to pneumococcal vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Mothers from 18 to 14 years of age in the third trimester of pregnancy,
* with normal medical and obstetric history,
* who plan to deliver their infant in Dhaka city and remain there for 12m

Exclusion Criteria:

* Maternal history of systemic disease,
* Maternal history of previous complicated pregnancies, preterm delivery, abortions, or birth with congenital anomalies.
* Maternal hypersensitivity to any vaccination, or
* Maternal receipt of pneumococcal vaccine in the last 3 years.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 680
Dates: Start 2004-08; Study Completion 2006-12

PRIMARY OUTCOMES:
Serum anti pneumococcal polysaccharide IgG antibody at 20 weeks of age
local and systemic reactions within 2 weeks of vaccination

SECONDARY OUTCOMES:
Level and duration of serum IgG antibody to pneumococcus up to 1 year of age.

CONTACTS AND LOCATIONS:
Overall Officials: M C Steinhoff, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- ICDDRB, Dhaka, Bangladesh

REFERENCES:
- [Derived] Schlaudecker EP, Steinhoff MC, Omer SB, McNeal MM, Roy E, Arifeen SE, Dodd CN, Raqib R, Breiman RF, Zaman K. IgA and neutralizing antibodies to influenza a virus in human milk: a randomized trial of antenatal influenza immunization. PLoS One. 2013 Aug 14;8(8):e70867. doi: 10.1371/journal.pone.0070867. eCollection 2013. PMID 23967126
- [Derived] Omer SB, Zaman K, Roy E, Arifeen SE, Raqib R, Noory L, Seib K, Breiman RF, Steinhoff MC. Combined effects of antenatal receipt of influenza vaccine by mothers and pneumococcal conjugate vaccine receipt by infants: results from a randomized, blinded, controlled trial. J Infect Dis. 2013 Apr;207(7):1144-7. doi: 10.1093/infdis/jit003. Epub 2013 Jan 8. PMID 23300160
- [Derived] Steinhoff MC, Omer SB, Roy E, El Arifeen S, Raqib R, Dodd C, Breiman RF, Zaman K. Neonatal outcomes after influenza immunization during pregnancy: a randomized controlled trial. CMAJ. 2012 Apr 3;184(6):645-53. doi: 10.1503/cmaj.110754. Epub 2012 Feb 21. PMID 22353593
- [Derived] Zaman K, Roy E, Arifeen SE, Rahman M, Raqib R, Wilson E, Omer SB, Shahid NS, Breiman RF, Steinhoff MC. Effectiveness of maternal influenza immunization in mothers and infants. N Engl J Med. 2008 Oct 9;359(15):1555-64. doi: 10.1056/NEJMoa0708630. Epub 2008 Sep 17. PMID 18799552